CLINICAL TRIAL: NCT02669251
Title: A Phase 1b/2 Study of Alvelestat (MPH966), an Oral Neutrophil Elastase Inhibitor, in Bronchiolitis Obliterans Syndrome After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Alvelestat (MPH966), an Oral Neutrophil Elastase Inhibitor, in Bronchiolitis Obliterans Syndrome After Allogeneic Hematopoietic Stem Cell Transplantation
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 160060; 16-C-0060
Record Dates: First submitted 2016-01-29; First posted 2016-02-01 (Estimated); Last update posted 2025-12-09 (Actual); Status verified 2025-12-05

CONDITIONS: Chronic Graft vs Host Disease; Chronic Graft-Versus-Host Disease; Bronchiolitis Obliterans Syndrome
Keywords: Optimal Biologic Dose; Safety; Chronic Graft-Versus-Host Disease (cGVHD); Inflammatory Lung Disease; FEV1
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1b (Experimental): Phase Ib dose escalation
  Interventions: Drug: MPH966
- Phase 2 (Experimental): MTD po bid on days 1-28
  Interventions: Drug: MPH966

INTERVENTIONS:
Drug: MPH966 — Phase 1b Cycle= 14 days: Each dose level will increase by 60mg PO BID, up to a maximum of 240mg PO BID
  Phase 2 Cycle=28 days: MTD PO BID

SUMMARY:
Background:

Bronchiolitis obliterans syndrome (BOS) is a complication people can experience after hematopoietic stem cell transplant. It usually affects people with chronic graft versus host disease (cGVHD). This occurs when donor stem cells attack the cells of the person who received them. BOS reduces airflow and oxygen levels in the body. It may be caused by neutrophil elastase in the body. Researchers believe the new drug alvelestat (MPH966) may help.

Objectives:

To test the safety of alvelestat (MPH966) and see what dose best inhibits neutrophil elastase in people with BOS after a stem cell transplant. To study how well the best dose improves lung function in those people.

Eligibility:

Adults 18 and older who have had a hematopoietic stem cell transplant and have cGVHD and BOS.

Design:

Participants will be screened with a medical history, physical exam, and blood and urine tests. They will have lung function and heart function tests. They will have computed tomography scans of the chest.

Study part 1: Participants will take the starting dose of the study drug by mouth twice a day for 14 days. This is 1 cycle. They will get different doses, for up to 4 cycles.

Study part 2: Participants will take the study drug twice a day by mouth at the dose set in part 1, for up to 12 months.

Participants will keep medicine diaries.

Participants will have several study visits. These may include:

Repeats of the screening tests.

Bronchoscopy with bronchoalveolar lavage.

Sputum samples taken.

6-minute walking test.

cGVHD assessment and answer questions.

Participants will be contacted after the study for up to 24 months.

DETAILED DESCRIPTION:
Background:

* Chronic graft-versus-host disease (cGVHD) is the leading cause of non-relapse morbidity and mortality in persons after allogeneic hematopoietic stem cell transplantation (SCT).
* Bronchiolitis obliterans syndrome (BOS) is a complication of cGVHD associated with a high morbidity and mortality, and treatment options are limited.
* Neutrophil elastase (NE) is a protease released by neutrophils in the setting of inflammation, and has been implicated in the pathogenesis of BOS.
* Alvelestat (MPH966) (Formerly known as AZD9668) is a potent and selective inhibitor of NE that has demonstrated evidence of target inhibition and a good safety profile in patients with inflammatory lung diseases, but has not been evaluated in BOS.

Objectives:

Phase 1b:

To determine the optimal biologic dose (OBD) based on maximal NE inhibition measured in blood, and to determine the safety of alvelestat (MPH966) in patients with BOS after SCT

Phase 2:

To determine the clinical efficacy of alvelestat (MPH966) at the OBD in patients with BOS after SCT, based on the proportion of patients with stable or improved forced expiratory volume in 1 second (FEV1) on pulmonary function testing

Eligibility:

Inclusion criteria:

* Age >=18 years
* BOS after SCT and moderate to severe cGVHD as defined by the NIH consensus criteria
* Within 5 years from the time of diagnosis (Phase 2 only)
* Karnofsky performance status >= 60%
* If on systemic cGVHD therapy, must be receiving stable or tapering doses in the preceding 4 weeks
* Patients will be required to have received prior treatment with a regimen consisting of inhaled steroids and montelukast +/- azithromycin for at least 3 months prior to enrollment, unless there is evidence of progression or unsatisfactory response while on this regimen prior to 3 months of treatment, as deemed by the treating or referring physician.
* Patients who are on azithromycin, an antibiotic used in the treatment of BOS, will need to discontinue for at least 2 weeks prior to enrollment

Exclusion criteria:

* FEV1 < 30% (based on absolute percent predicted using USA-ITS-NIH equation) on pulmonary function testing
* Prior use of neutrophil elastase inhibitors
* Progressive malignancy
* Uncontrolled infection or any major organ dysfunction as defined by the protocol

Design:

Phase 1b:

* This is a Phase 1b trial to determine the OBD and safety of alvelestat (MPH966) in patients with BOS after SCT.
* This trial will use an intra-patient dose escalation schedule. The starting dose will be 60mg twice daily for 2 weeks, and the dose will be increased by 60mg with each escalation every 2 weeks until a maximum dose of 240mg twice daily is reached for a total treatment period of 8 weeks. After completion of the dose escalation phase, patients will have the option to continue the dose at which maximal NE inhibition and safety are demonstrated for up to 6 additional months.
* The co-primary endpoint of OBD will be defined as the dose level at which the maximal NE inhibition occurs, and at which no more than 1/3 of patients experience a DLT. NE activity will be measured in the blood at baseline and with each dose escalation, and will be compared between dose levels to determine the OBD.
* The co-primary endpoint of safety will be determined by monitoring adverse events and dose limiting toxicities (DLT) as defined by the protocol. Further dose escalation will cease in a patient who experiences a DLT. In addition, no subsequent patients will be treated at or beyond the dose in which 1/3 of patients have experienced a DLT.
* A total of 10 patients will be enrolled in the Phase 1b trial.

Phase 2:

* This is a Phase 2 trial to determine the efficacy of alvelestat (MPH966) at the OBD in patients with BOS after SCT, as measured by stabilization or improvement of FEV1 (based on absolute percent predicted) after 6 months of treatment.
* Patients will receive alvelestat (MPH966) using an intra-patient dose escalation schedule. The starting dose will be 60 mg twice daily for 2 weeks, and the dose will be increased by 60 mg twice daily with each dose escalation every 2 weeks until a maximum dose of

  240 mg twice daily is reached for a total treatment period of 18 weeks (total of 6 cycles). There is an optional continuation phase for 24 more weeks (cycles 7-12) with each cycle being 28 days and pulmonary function testing with measurement of FEV1 will be performed to determine the primary endpoint.
* Response assessments will occur every 3 months with primary efficacy endpoint evaluated at 6 months. Patients with stable or responding disease will have the option to continue therapy for another 6 months.
* As an early stopping rule for futility, if 0-2 of the first 8 patients enrolled have responded, then no further patients will be accrued. A total of 20 patients may be needed for evaluation in phase II.

In order to allow for a small number of inevaluable patients, the accrual ceiling will be set at 34 patients across both phases.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have undergone hematopoietic stem cell transplantation and have moderate to severe chronic GVHD as defined by the NIH consensus criteria.
* Patients must have BOS as defined by either of the two following criteria (A or B):

(A) BOS per NIH consensus criteria (2014 updated criteria). To meet the criteria for BOS, all of the following must be present, in addition to at least one distinctive manifestation of cGVHD:

* FEV1/vital capacity <0.7 or the fifth percentile of predicted
* FEV1 <75% of predicted with >= 10% decline over less than 2 years. FEV1 should not correct to >75% with albuterol
* Absence of infection in the respiratory tract
* One of the 2 supporting features of BOS:

  1. Evidence of air trapping by expiratory CT or small airway thickening or bronchiectasis by high-resolution CT, or
  2. Evidence of air trapping by PFTs: residual volume >120% predicted or residual volume/total lung capacity elevated outside the 90% confidence interval.

If a patient carries the diagnosis of cGVHD by virtue of organ involvement elsewhere, then only the first 3 criteria above are necessary.

(B) BOS, expanded NIH criteria

* FEV1/vital capacity >0.7
* FEV1 <75% of predicted with >= 10% decline over less than 2 years. FEV1 should not correct to >75% with albuterol
* Absence of infection in the respiratory tract
* One of the supporting features of BOS:

  1. Evidence of air trapping by expiratory CT
  2. small airway thickening or bronchiectasis by high-resolution CT
  3. Evidence of air trapping by PFTs: residual volume >120% predicted or residual volume/total lung capacity elevated outside the 90% confidence interval.

     * For the Phase 1b study, patients may have had the diagnosis of BOS for any period of time. For the Phase 2 study, patients must be within 5 years from the time of diagnosis. Patients may be at any time interval after SCT as long as the criteria for chronic GVHD and BOS are met.
     * If patients are taking systemic therapy for cGVHD at the time of enrollment, they must be receiving stable or tapering doses within the previous 4 weeks. Patients are not required to have completed a course of steroids prior to enrollment.
     * Age >=18 years.
     * Karnofsky >=60%
     * Patients must have adequate organ and marrow function as defined below:
* Leukocytes >=3,000/mcL
* Absolute neutrophil count >=1,000/mcL
* Platelets >=50,000/mcL
* Total bilirubin <=3 x institutional upper limit of normal, unless there is a known history of Gilbert's disease
* AST(SGOT)/ALT(SGPT) <=2 x institutional upper limit of normal
* Serum creatinine <=1.5 mg/dL OR Creatinine clearance >=60 mL/min as estimated by GFR per DLM standards

  * Patients will be required to have received prior treatment with a regimen consisting of inhaled steroids and montelukast +/- azithromycin for at least 3 months prior to enrollment, unless there is evidence of progression or unsatisfactory response while on this regimen prior to 3 months of treatment, as deemed by the treating or referring physician. Patients who are on azithromycin will need to discontinue for at least 2 weeks prior to enrollment.
  * Agree to adhere to methods of contraception and other fertility control measures:

The effects of alvelestat (MPH966)on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study therapy. Contraception should be used up until 1 week of discontinuing study medication.

-Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* FEV1 <30% (based on absolute percent predicted using USA-ITS-NIH equation) on pulmonary function testing
* Patients with clinically relevant abnormal ECG findings, including abnormal QTc>500 ms on screening ECG (Note: If a patient has a QTc interval >500 ms on screening ECG, the screening ECG may be repeated twice [at least 24 hours apart] for a total of 3 ECGs).
* Patients who are receiving any other investigational agents
* Recurrent or progressive malignancy requiring anticancer treatment
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, acute kidney injury, or psychiatric illness/social situations within the previous 4 weeks that would limit compliance with study requirements.
* Pregnant women are excluded from this study because the teratogenic effects of alvelestat (MPH966) are unknown. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with alvelestat (MPH966), nursing should be discontinued if the mother is treated with this agent.
* Prior use of neutrophil elastase inhibitors
* Patients with a history of cirrhosis, esophageal varices, ascites and hepatic encephalopathy
* History of other chronic diseases (i.e., metabolic associated steatohepatitis (MASH), autoimmune hepatitis, primary biliary cholangitis, primary sclerosing cholangitis, Wilson's disease, haemochromatosis)
* Patients with a history of significant alcohol consumption for a period of more than 3 consecutive months within 1 year prior to screening. NOTE: Patients must also be willing to refrain from drinking alcohol during study participation, until end of study drug administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-04-28 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Optimal biologic dose (OBD) based on maximal NE inhibition measured in sputum | 8 weeks after study drug initiation
  Dose-finding.
To determine the clinical efficacy of MPH966 at the OBD in patients with BOS after SCT | 6 months
  Efficacy.
determine the safety of MPH966 | 8 weeks after study drug initiation
  Safety.

SECONDARY OUTCOMES:
Phase 1b and 2: Pharmacokinetics of blood and sputum | Phase 1b: Baseline, first day of each cycle at dose escalation. Phase 2: Baseline, C1D1, C3D1, C6D1.
  Pharmacokinetics of study drug.
Phase 1B: Correlation of NE activity in blood with sputum measurements | Phase 1b: Pre/post dose on day 1 of each dose level and at start of continuation phase. Phase 2: Pre/post dose on day one of each dose level.
  Efficacy/drug effect on laboratory values.
Phase 1B and 2: Determine the impact on lung inflammatory markers based on levels in blood, sputum and BAL fluid | Phase 1b: Baseline, 8 wees. Phase 2: Baseline, 3 months and 6 months (end of treatment).
  Efficacy/drug effect on laboratory values.
Phase 2: Efficacy testing via NIH Lung Symptom Score, 6 minute walk test, survival, FEV1 slope measured from baseline, and other PFT measurements | Baseline, C1D1, D4D1, C7D1, c10D1, Off treatment.
  Efficacy.
Phase 1B and 2: Determine effect on patient-reported outcomes viaLee cGVHD Symptom Scale, HAP, FACT-BMT | Phase 1B: C1D1, D1 of continuation phase, D1 of Cycle 11+, Off treatment. Phase 2: Baseline, D1 of C7-12, Off treatment.
  Analysis of patient-reported outcomes.
Phase 2: Determine effect on markers of target inhibition in sputum and blood | Baseline, 3 months and 6 months (end of treatment) or off study.
  Efficacy/drug effect on laboratory values.

CONTACTS AND LOCATIONS:
Overall Officials: Najla El Jurdi, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-C-0060.html